CLINICAL TRIAL: NCT00529334
Title: A Pilot Study of CyberKnife Radiosurgery Delivered to the Partial Breast for Women With Stage 0, 1, or IIA (<=3cm) Breast Cancer
Brief Title: A Pilot Study of CyberKnife Radiosurgery Delivered to the Partial Breast
Acronym: CK-PBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Georgetown University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUMC 2007-153
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Partial breast irradiation; Radiosurgery; CyberKnife; Radiotherapy; PBI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): CyberKnife Partial Breast Irradiation (PBI)
  Interventions: Radiation: CyberKnife Partial Breast Irradiation

INTERVENTIONS:
Radiation: CyberKnife Partial Breast Irradiation — Body radiosurgery will be delivered to the lumpectomy cavity with specified margin. Radiation dose will be 600 cGy x 5 stages = 3000 cGy over five to ten total days.

SUMMARY:
This pilot study will evaluate the technical feasibility and acute toxicity of Partial Breast Irradiation (PBI) with the CyberKnife in anticipation of a larger multi-institutional Phase II study. It will evaluate quality of life (QOL) issues as they relate to treatment related side effects, cosmetic result, and patient convenience.

Radiosurgery is defined as the stereotactic delivery of ionizing radiation in 5 stages or less to a designated target with sub-millimeter accuracy. Radiosurgery in the context of this protocol will be given to the region of the tumor bed within 7 weeks of lumpectomy and sentinel/axillary node sampling over a period of five to ten days using the CyberKnife (CK). Subjects will receive CK before chemotherapy, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* DCIS or infiltrating ductal carcinoma of the breast <= 3cm
* margins clear by at least 2 mm
* age >=45 years

Exclusion Criteria:

* invasive lobular carcinoma
* multicentric disease
* nodal metastases
* breast implants
* pregnancy
* connective tissue disease

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
1. To evaluate the feasibility of CyberKnife body radiosurgery as the sole radiation therapy for this patient population 2. To evaluate the complication rate of CyberKnife body radiosurgery as the sole radiation therapy for this patient population | 1 year

SECONDARY OUTCOMES:
1. To evaluate the local control rate of CyberKnife body radiosurgery as the sole radiation therapy for this patient population. 2. To evaluate Quality of Life after CyberKnife body radiosurgery PBI. | 1 - 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson EC Moulds, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgtown University Medical Center, Washington D.C., District of Columbia, United States